CLINICAL TRIAL: NCT00913445
Title: Wound Healing and Cosmetic Result After Emergency Appendicectomy in Adult Patients: a Prospective, Randomised Trial Comparing Two Methods of Wound Closure
Brief Title: Wound Healing After Emergency Appendicectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Tuomo Rantanen MD,PhD, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R09060
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-05

CONDITIONS: Appendicitis
Keywords: Appendicitis; appendicectomy; stitches; wound healing; cosmetic results
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgery, absorbable stitches (Active Comparator): wound healing after absorbable and nonabsorbable stitches are compared
  Interventions: Procedure: appendicectomy
- surgery, nonabsorbable stitches (Active Comparator)
  Interventions: Procedure: appendicectomy

INTERVENTIONS:
Procedure: appendicectomy — Wound healing after absorbable and nonabsorbable stitches are compared

SUMMARY:
The purpose of this trial is to compare two techniques of wound closure in open appendicectomies in adult patients: continuous, absorbable, intradermal suture and interrupted, non-absorbable sutures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with acute appendicitis

Exclusion Criteria:

* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Wound heeling | 14 days after operation

SECONDARY OUTCOMES:
Cosmetic result | 1 year after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland